CLINICAL TRIAL: NCT07290400
Title: Phase 2 Crossover Study Assessing the Effect of Moderate Alcohol Intake on the Absorption and Onset of Action of Hezkue® Sildenafil Oral Suspension
Brief Title: Effect of Moderate Alcohol on Absorption and Onset of Hezkue Sildenafil Suspension
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aspargo Labs, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASP-022-Sil
Record Dates: First submitted 2025-12-11; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-Arm Crossover (Experimental)
  Interventions: Drug: Hezkue Sildenafil Oral Suspension
- Hezkue® With Moderate Alcohol Intake (Experimental): Participants will receive Hezkue® sildenafil oral suspension administered following standardized moderate alcohol intake in one study period. Pharmacokinetic, absorption, onset of action, and safety assessments will be conducted following dosing.
  Interventions: Drug: Hezkue Sildenafil Oral Suspension; Other: Moderate Alcohol Intake

INTERVENTIONS:
Drug: Hezkue Sildenafil Oral Suspension — Hezkue® sildenafil oral suspension will be administered as a single oral dose in each study period under different alcohol intake conditions (such as with and without moderate alcohol consumption), according to the randomized crossover design. Pharmacokinetic, absorption, onset of action, and safety parameters will be assessed after each administration.
Other: Moderate Alcohol Intake — A standardized moderate amount of alcohol will be administered under controlled conditions prior to dosing with Hezkue® sildenafil oral suspension in designated study periods, according to the protocol-defined alcohol intake procedures.
  Arms: Hezkue® With Moderate Alcohol Intake

SUMMARY:
This is a Phase 2, open-label, randomized crossover study assessing the effect of moderate alcohol intake on the absorption and onset of action of Hezkue® sildenafil oral suspension in adult subjects. Participants will receive Hezkue® under different alcohol intake conditions in randomized sequence. Pharmacokinetic sampling and onset assessments will be performed after each administration, and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male adults 21 to 65 years of age, inclusive
* Documented history of erectile dysfunction for at least 6 months, as determined by the investigator
* In a stable sexual relationship and willing to attempt sexual activity as required by study procedures, if applicable
* Medically stable based on medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations, in the opinion of the investigator
* Able, in the investigator's judgment, to safely consume moderate amounts of alcohol as defined in the protocol
* Willing to abstain from alcohol outside of protocol-specified intake during the study
* Able to understand and provide written informed consent before any study-specific procedures are performed
* Willing and able to comply with all study procedures, including dosing, washout periods, pharmacokinetic sampling, onset assessments, and safety monitoring

Exclusion Criteria:

* Known hypersensitivity or contraindication to sildenafil, other PDE5 inhibitors, alcohol, or any component of the Hezkue® formulation
* Use of nitrates, nitric oxide donors, guanylate cyclase stimulators (such as riociguat), or other prohibited medications within a protocol-defined period
* Clinically significant cardiovascular disease, including coronary artery disease, heart failure, clinically important arrhythmias, recent stroke, or uncontrolled hypertension or hypotension
* Resting blood pressure or heart rate outside protocol-defined acceptable ranges at screening or baseline, in the opinion of the investigator
* Significant hepatic, renal, neurologic, psychiatric, endocrine, hematologic, or respiratory disease that could increase risk or interfere with study assessments
* History of syncope, significant orthostatic hypotension, or other conditions that may be worsened by sildenafil or alcohol
* History of alcohol use disorder, binge drinking, or other substance use disorder, as determined by the investigator
* Positive urine drug screen or positive alcohol test at screening or admission (outside protocol-specified alcohol administration)
* Use of prescription or over-the-counter medications, herbal products, or dietary supplements within 14 days before first dosing unless approved by the investigator
* Positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV
* Participation in another clinical study or receipt of an investigational product within 30 days or 5 half-lives, whichever is longer
* Donation of 450 mL or more of blood, or significant blood loss, within 8 weeks before first dosing
* Any condition or circumstance that, in the opinion of the investigator, would make the participant unsuitable or interfere with study conduct or interpretation

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Time to Onset of Effect as Assessed by Participant-Reported Erectile Response | From dosing up to approximately 4 hours postdose in each study period
Area Under the Plasma Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC₀-t) of Sildenafi | From predose up to approximately 24 hours postdose in each study period

IPD SHARING:
Plan to Share IPD: No